CLINICAL TRIAL: NCT00524095
Title: Bronchiectasis in COPD Patients : Role of Prophylaxis With Inhaled Steroids and Antibiotic on the Natural History of the Disease
Brief Title: Bronchiectasis in Chronic Obstructive Pulmonary Disease (COPD) Patients: Role of Prophylaxis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: we decided not to go on treatment phase
Sponsor: University of Milan (Other)
Responsible Party: Francesco Blasi, University of Milan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRIN2005; MIUR 2005067041 PRIN 2005
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Bronchiectasis; Pulmonary Disease; Chronic Bronchitis
Keywords: prophylaxis; Antibiotic; inhaled steroids; bronchiectasis; prevalence; chronic bronchitis
MeSH Terms: conditions — Bronchiectasis; Lung Diseases; Bronchitis, Chronic | interventions — Azithromycin; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): standard of care
- 2 (Experimental): azithromycin 500 mg once a day three times a week for 6 months and then inhaled steroids (fluticasone 500 ug bid) for 6 months
  Interventions: Drug: azithromycin and fluticasone
- 3 (Experimental): inhaled steroids (fluticasone 500 ug bid) for 6 months and then azithromycin 500 mg once a day three times a week for 6 months
  Interventions: Drug: fluticasone and azithromycin

INTERVENTIONS:
Drug: azithromycin and fluticasone — azithromycin 500 mg once a day three times a week for 6 months and then inhaled steroids (fluticasone 500 ug bid) for 6 months
  Other Names: azithromycin; fluticasone
  Arms: 2
Drug: fluticasone and azithromycin — inhaled steroids (fluticasone 500 ug bid) for 6 months and then azithromycin 500 mg once a day three times a week for 6 months
  Other Names: fluticasone; azithromycin
  Arms: 3

SUMMARY:
Bronchiectasis is a chronic pulmonary disease characterized by an irreversible dilatation of the bronchi. The current view of the pathogenesis of bronchiectasis considers initial colonization of the lower respiratory tract by different microorganisms as the first step leading to an inflammatory response characterized by neutrophil migration within the airways and secondary secretion of a variety of tissue-damaging oxidants and enzymes such as neutrophil elastase and myeloperoxidase. Persistence of microorganisms in the airways because of impairment in mucus clearance may lead to a vicious circle of events characterized by chronic bacterial colonization, persistent inflammatory reaction, and progressive tissue damage. The exact prevalence of bronchiectasis in COPD patients is not known. It would be important to assess the prevalence, the kind of bronchiectasis and the bacterial colonisation. These are all important features that can be related to the natural history of COPD and to the therapeutic management of patient with COPD and bronchiectasis. Recent data indicate that macrolide long-term treatment and inhaled steroids therapy are both associated with a reduced rate of exacerbation, bronchial colonization and inflammation The present study will address, on a relatively large number of patients, the prevalence of bronchiectasis in COPD subjects using a multislice CT scan technique applied in all the units and centrally analysed by Unit 2 and 4. This analysis will determine the presence and the morphology of bronchiectasis. Bacterial colonization and inflammatory parameters will be evaluated on blood and exhalate bronchial condensate. Concerning bacterial colonization molecular biology techniques (Qualitative PCR and quantitative real time PCR) will be applied. ELISPOT technique for the evaluation of specific immune response will be used.Electron and optical microscopy techniques will be applied on bronchial biopsy samples obtained in a subgroup of patients enrolled. During the second study year, a randomized trial on patients with bronchiectasis will be performed. Patients will be randomized to receive a macrolide or inhaled steroids or standard of care for 6 months with a follow-up of 6 months. All the inflammatory, microbiologic and functional parameters described above will be recorded. A clinical and functional evaluation will be applied looking to number of exacerbations, quality of life, respiratory function parameters.

DETAILED DESCRIPTION:
AIMS OF THE STUDY

As previously described the research program aims are the following:

* definition of bronchiectasis prevalence in patients affected by chronic obstructive pulmonary disease.
* After bronchiectasis patients identification, we will evaluate the pathophysiologic implications, and microbiologic and inflammatory features of this subgroup in comparison to non-bronchiectasis patients.
* Finally, the research will address the effects of long-term treatments with inhaled steroids and antibiotic on the natural history of the disease and their pathophysiologic implications. To these purposes, the study will be divided into two sections. In the Ist section 400 patients with COPD will be recruited. In these patients we intend to assess the prevalence of bronchiectasis using a CT spiral scanning. We will also detect bacterial colonisation by real time PCR and ELIspot technique, and airway inflammation by a non-invasive method (exhaled breath condensate) comparing patients with and without bronchiectasis.

COPD patients with bronchiectasis:

In this population we will study the effect of different "prophylaxis" i.e., macrolide and inhaled steroids.

Details of the Interventions Proposed STABLE COPD The patient will attend the clinic in the morning for enrolment, and provide written informed consent. During the visit medical history will be recorded and subjects will undergo a physical examination and lung function testing at baseline and post salbutamol 200 mcg. CT scan, exhaled breath condensate and the venopuncture will also be performed. Sputum samples will be obtained for bacterial colonization assessment.

Respiratory Assessment:

Lung function testing will be performed using a Fleish No. 3 heated pneumotachograph; the plethysmographic measurements, thoracic gas volume (TGV), residual volume (RV), total lung capacity (TLC), will be assessed using a body plethysmograph (Werner Gut, Basle, Switzerland) with electronic BTPS compensation at a constant volume (850L). DLCO determination will be performed.

CT scan All the multislice CT (MSCT) scan performed will be centrally analysed by UO 4 . The following protocol will be followed

1. MSCT in inspiration at TLC with slice of 1 mm every 10 + 3 expiratory slices at RV using three predetermined levels (aortic arch, tracheal carina, right basal common vein)
2. Technical parameters: 120 kV, 220 mA, filter bone, FOV including both lung, lung parenchyma window (-600/1600 HU)
3. All CT will be saved on CD rom Two radiologists will analyse the same CT, every discrepancy will be solved by consensus

The diagnosis and evaluation of bronchiectasis will be performed according to Webb et al. (1):

The evaluation will be performed lobe by lobe including lingula (total lobes= 6)

1. bronchiectasis extension on lobar base: 0, 1 (< 25% of the lobe), 2 (25-50%), 3 (>50%) - MAX TOT 18
2. severity and kind of bronchiectasis and semi-quantitative, comparing the diameter to that of the adjacent artery: 0, 1 (bronchial diameter equal to 100-200% artery diameter), 2 (200-300%), 3 (> 300%) - MAX TOT 18
3. Thickness of bronchial walls: 0, 1 (Thickness < 50% artery diameter), 2 (50-100%), 3 ( complete obliteration of lumen or Hydro-air levels) - MAX TOT 18
4. Evaluation of emphysema (visual score on three levels (inspiration) (aortic arch, carina, vein)
5. Evaluation of air trapping in expiration (idem)
6. Bullae
7. Ground glass areas (extension by visual score)
8. bronchiolitis: prevalent site, lobar involvement, severity ( 0,1,2,3)
9. Pulmonary artery diameter (pathological if > 2,9 cm)
10. Other features

Exhaled breath condensate:

Exhaled breath condensate will be collected by using a condenser, which allows the non-invasive collection of nongaseous components of the expiratory air (EcoScreen, Jaeger, Germany). Subjects breathe tidally through a mouthpiece connected to the inlet for 8 min while wearing a nose-clip. The mouthpiece is also used as a saliva trap. Approximately 1 ml of breath condensate is collected and stored at -70° C. IL-6, IL-8, TNF-a and cysteinyl-leukotrienes (cys-LTs) will be measured by specific enzyme immunoassays (EIA) (Cayman Chemical, Ann Arbor, MI). Moreover proteomic analysis will be performed on the subset of patients enrolled by UO1 as previously reported (2); briefly, one-dimensional and two-dimensional electrophoresis will be performed and for qualitative evaluation and mass spectrometry analysis, the gels will be stained with silver nitrate, with or without glutaraldehyde in the sensitization step and formaldehyde in the impregnation solution. Spot volumes will be calculated using Image J 1.29x (W. Rasband, National Institutes of Health, Bethesda, Maryland) for one-dimensional gels, and with PDQUEST (Biorad, Hercules, California) for two-dimensional gels.

Serum Samples:

Serum aliquots will be arranged in duplicate and stored at - 20°C until the time of analysis. IL-6, IL-8, TNF-a and cysteinyl-leukotrienes (cys-LTs) will be measured by specific enzyme immunoassays (EIA) (Cayman Chemical, Ann Arbor, MI).

C-reactive protein and procalcitonin will be also measured.(3) UO 1 The ex-vivo Enzyme-Linked ImmunoSPOT (ELISPOT) assay is the most sensitive tool to detect and quantify the antigen-specific T-cell response, and can detect and enumerate T-cells producing one or more cytokines in response to specific antigens. This technique has been already used to detect low numbers of antigen-specific T-cells in infectious disorders, with particular emphasis to intracellular pathogens such as Mycobacterium tuberculosis . The ELISPOT technique is becoming a standard reference for the monitoring of many infectious diseases, including HIV infection, and is becoming more and more used in advanced clinical immunological applications, such as the detection of an antigen-specific T cell immune responses to oncogene peptides.

In the context of the proposed project, the ELISPOT technology will be used to detect the presence of a systemic (blood) and local (bronchoalveolar lavage) antigen-specific response using peptide pools of non tuberculous mycobacteria and other intracellular bacteria (such as Mycoplasma pneumoniae), bacteria (such as Pseudomonas spp) and fungi (such as Aspergillus species). The ELISPOT tests will be performed on samples of whole blood (after Ficoll separation of peripheral mononuclear cells) and bronchoalveolar cells measuring the number of T cells producing interferon-gamma after an overnight incubation with the specific antigenic peptide pools. (4-8)

Sputum collection:

A sample of spontaneous sputum will be obtained from all patients. Alternatively induced sputum according to Pizzichini, et al (9) will be collected. In summary, induced sputum is obtained after inhalation of hypertonic saline water at 3% for 20 minutes using an ultrasonic nebulizer (Ultraneb 2000; DeVilbiss Healthcare Inc, Somerset, PS, USA).Only samples of sputum degree IV or V of Murray-Washington classification (10) will be processed. A sputum sample will be frozen at -70°C for bacterial DNA detection using a PCR (qualitative analysis) and real time PCR (quantitative analysis) techniques.

The following Bacteria wil be detected using standard protocol in use in UO1: H. influenzae, M. catarrhalis, S. pneumoniae, P.

aeruginosa, Mycoplasma pneumoniae, Chlamydia pneumoniae. An aliquot will be cultivated using standard microbiologic techniques Patients 400 patients will be recruited at the UO 1,2,3 e 5. All the CT scan will be collected and examined at UO 4. UO2 will serve as second observer in a double-blind fashion; any discrepancy will be solved by consensus.

One subgroup of patients with stable COPD (n=15) and an subgroup of patients with COPD and bronchiectasis (n=15) will undergo bronchoscopy with biopsy collection. Subjects will be premedicated with atropine and anesthetized topically with lidocaine.

Bronchoscopy will be performed with a flexible fiberoptic bronchoscope. Bronchial biopsies will be taken through the bronchoscope with standard forceps from the carina of the basal segment bronchus of the right lower lobe. From this area two specimens will be obtained in each patients. Bronchial biopsies obtained will be prepared for electronic and light microscopy analysis (UO3 and UO 1).

Sample size: we can expect at least a 30% prevalence of bronchiectasis that means 120 patients to be included in the second step of the study (11)

COPD PATIENTS WITH BRONCHIECTASIS:

In this population we will study the effect of different "prophylaxis" i.e. macrolide and inhaled steroids. The population will be followed for 12 months.

The following procedure will be performed every 3 months and at each exacerbations:

Clinical assessment, Exhaled breath condensate, Serum Sampling, Sputum collection.

On biological samples all the previously described techniques plus renal and hepatic function tests (safety) will be performed.

Sputum culture will be performed to assess bacterial flora and resistance patterns.

Design of the study:

120 patients will be randomized in 3 groups (40 pts) to receive :

1. Standard of care
2. azithromycin 500 mg OD 3 days a week (Monday, Wednesday, Friday) for 6 months and then inhaled steroids (fluticasone 500 ug bid) for 6 months
3. inhaled steroids (fluticasone 500 ug bid) for 6 months and then azithromycin 500 mg OD 3 days a week (Monday, Wednesday, Friday) for 6 months

End-points:

PRIMARY

* effects of treatments on bronchial inflammation parameters SECONDARY
* effects of treatments on exacerbations frequency
* effects of treatments on pulmonary function

Sample size:

We can expect a 40% difference between treated and non-treated patients for at least one among TNFa, IL6, IL8, and cysteinyl-leukotrienes. In this case we need 35 treated patients (for each arm) and 35 non-treated patients for an alpha error of 0.05 and a beta of 0.1.

ELIGIBILITY:
Inclusion Criteria:

* Smokers or former smokers of at least 10 pack-years
* COPD demonstrated by forced spirometry with FEV1 > 0,7 L, FEV1 post-BD <60% and FEV1/FVC < 70%
* Bronchodilator test performed at inclusion or no more than 6 months before inclusion should have been negative (increase in FEV1 < 200 ml and 12%, 10 minutes after administration of 2 puffs of salbutamol
* Stable phase defined by clinical criteria of the attending investigator, but at least 6 weeks from the last exacerbation
* Informed consent

Exclusion Criteria:

* Patients receiving oral corticosteroids at any dose or another immunosuppressor
* Formal contraindication for sputum collection or impossibility to obtain a sample of sputum valid for analysis.
* Allergy to steroids or macrolides

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
effects of treatments on bronchial inflammation parameters | six months

SECONDARY OUTCOMES:
effects of treatments on exacerbations frequency | six months
effects of treatments on pulmonary function | six months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Blasi, MD, Study Director — University of Milan Italy
Locations (4):
- Italy (4):
  - Istituto Malattie Respiratorie University of Milan, Milan
  - Clinica di Malattie dell'Apparato Respiratorio Università di Modena e Reggio Emilia, Modena
  - Dip. SCIENZE CARDIOLOGICHE, TORACICHE E VASCOLARI UNIVERSITY OF PADOVA, Padua
  - Dip. SCIENZE CLINICHE Università degli Studi di PARMA, Parma

REFERENCES:
- See also: official website of the Italian Ministry of Research and University (MUR) — http://www.ricercaitaliana.it/prin/dettaglio_prin-2005067041.htm